CLINICAL TRIAL: NCT06436768
Title: Effectiveness of Sugammadex Versus Neostigmine on the Reversal of Rocuronium-induced Neuromuscular Blockade in Patients With Myasthenia Gravis After Thoracoscopic Thymectomy: A Multicenter Randomized Controlled Trial
Brief Title: Efficacy and Safety of Sugammadex in Thoracoscopy Thymectomy for Chinese Adults With Myasthenia Gravis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRRCKY202 l-009-GZ (2023)-003; 320.6750.2020-21-10 (Other Grant/Funding Number: Wu Jieping Medical Foundation)
Record Dates: First submitted 2024-05-14; First posted 2024-05-31 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-05

CONDITIONS: Reversal of Neuromuscular Blockade
Keywords: neuromuscular blockade; Sugammadex; Neostigmine; Myasthenia gravis; Postoperative Residual Curarization
MeSH Terms: conditions — Myasthenia Gravis; Delayed Emergence from Anesthesia | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Intervention Model Description: Randomized parallel controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The doctors making the follow-up assessment were unaware of the treatment received, and none of the doctors who administered the injections carried out the follow- up evaluations. Thus, both the patients and the assessing doctors were remained unaware of the treatment received throughout the trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sugammadex group (S group) (Experimental): After the last dose of rocuronium, at reappearance of T2, a dose of 2.0 mg/kg sugammadex was administered.
  Interventions: Drug: Sugammadex
- Neostigmine group (N group) (Active Comparator): After the last dose of rocuronium, at reappearance of T2, a dose of 50 ug/kg neostigmine plus atropine 0.02 mg/kg was administered.
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — After the last dose of rocuronium, at reappearance of T2, a dose of 2.0 mg/kg sugammadex was administered.
  Dose will be according to participant actual body weight.
  Other Names: S group
  Arms: Sugammadex group (S group)
Drug: Neostigmine — After the last dose of rocuronium, at reappearance of T2, a dose of 50 ug/kg neostigmine (up to 5 mg maximum dose) plus atropine 0.02 mg/kg (up to 2 mg maximum dose) was administered.
  Dose will be according to participant actual body weight.
  Other Names: N group
  Arms: Neostigmine group (N group)

SUMMARY:
The purpose of this study was to demonstrate in patients with myasthenia gravis (MG) undergoing thoracoscopic thymectomy faster recovery from a moderate neuromuscular block induced by rocuronium after reversal at reappearance of T2 by 2.0 mg/kg sugammadex compared to 50 ug/kg neostigmine.

Methods: A total of 64 patients with MG undergoing thoracoscopic thymectomy will be randomly divided into two groups: Sugammadex group (S group) and Neostigmine group (N group). The same anesthesia methods will be applied in both groups. Patients of S group will receive a dose of 2.0 mg/kg sugammadex after the last dose of rocuronium, at reappearance of T2. Patients of N group will receive a dose of 50 ug/kg neostigmine after the last dose of rocuronium, at reappearance of T2. The primary endpoint is time from start of administration of sugammadex or neostigmine to recovery of train-of-four stimulation ratio (TOFr) to 0.9. Secondary end points include time from start of administration of sugammadex or neostigmine to recovery of TOFr to 0.8 and 0.7, time to extubation, clinical signs of neuromuscular recovery, hemodynamic changes after muscle relaxation antagonism, adverse effects, time to operating room (OR) discharge, time to post-anesthesia care unit (PACU) discharge, and pulmonary complications within 7 days after the operation.

DETAILED DESCRIPTION:
Due to neuromuscular transmission and functioning deficits, patients with myasthenia gravis (MG) are at increased risk of postoperative residual curarization (PORC), and may even develop into postoperative myasthenia crisis (PMC), which is a serious complication after thymectomy and increases the risk of death, with an incidence of up to 18.2%.

Effective reversal of neuromuscular blockade is crucial to ensure patient safety, reduce the incidence of PORC or PMC and prompt postoperative recovery. Traditionally, neostigmine, an acetylcholinesterase inhibitor, can be employed for neuromuscular blocking agent (NMBA) reversal. However, neostigmine is associated with potential drawbacks, such as delayed recovery and adverse muscarinic side effects.

Sugammadex, a selective relaxant binding agent, represents a relatively new alternative for NMBA reversal, specifically designed to encapsulate and inactivate aminosteroid NMBAs. The clinical benefits of sugammadex have been documented in several studies, demonstrating faster reversal of neuromuscular blockade and more predictable recovery profiles compared to neostigmine. However, the use of sugammadex in patients with MG remains an area of limited evidence. To date, to the best of our knowledge, there is a lack of prospective research to elucidate the application value of sugammadex in thymectomy in patients with MG.

This study is a prospective randomized controlled trial aimed at exploring the efficacy and safety of sugammadex compared to neostigmine for the reversal of neuromuscular blockade in patients with myasthenia gravis after thoracoscopic thymectomy.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with MG scheduled for elective thoracoscopic thymectomy

  * Aged 18 to 65 years
  * American society of Anesthesiologists (ASA) physical status classification system: I - III

Exclusion Criteria:

* Inability to obtain written informed consent
* With severe renal or hepatic dysfunction
* A plan to return to ICU with intubation postoperation
* A family history of malignant hyperthermia
* Suspected difficult airway
* Allergy to medications involved in the study
* A contraindication for neostigmine or sugammadex administration
* The patient's arm is not available for neuromuscular monitoring
* Patients receiving medication known to interfere with NMBAs (e.g., anticonvulsants, antibiotics, magnesium salts)
* Pregnant or lactating patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Recovery time | After operation within 24 hours
  The comparison of the recovery periods between groups when the start of administering reversal agent to the recovery of TOF ratio≥ 0.9

SECONDARY OUTCOMES:
Time from start of administration of sugammadex or neostigmine to the train-of-four stimulation ratio (TOFr) 0.8 | After operation within 120 minutes
  Muscle relaxation monitoring was performed with an accelero-myography (AMG) neuromuscular monitor by assessment of the TOF responses of adductor pollicis muscle to ulnar nerve stimulation every 15 seconds. T1 and T4 refer to the amplitudes of the first and fourth twitches, respectively, after TOF nerve stimulation. The TOFr, that is T4/T1 Ratio (expressed as a decimal of up to 1.0) represents the extent of recovery from neuromuscular blockade (NMB). A faster time to TOFr 0.8 indicates a faster recovery from NMB.
Time from start of administration of sugammadex or neostigmine to the train-of-four stimulation ratio (TOFr) 0.7. | After operation within 120 minutes
  Muscle relaxation monitoring was performed with an accelero-myography (AMG) neuromuscular monitor by assessment of the TOF responses of adductor pollicis muscle to ulnar nerve stimulation every 15 seconds. T1 and T4 refer to the amplitudes of the first and fourth twitches, respectively, after TOF nerve stimulation. The TOFr, that is T4/T1 Ratio (expressed as a decimal of up to 1.0) represents the extent of recovery from neuromuscular blockade (NMB). A faster time to TOFr 0.7 indicates a faster recovery from NMB.
Extubation time | After operation within 60 minutes
  The time period between administering a reversal agent to extubation
Time to discharge from the operating room | After operation within 60 minutes
  The time period between administering a reversal agent to operating room discharge
Time to discharge from recovery room | After operation within 120 minutes
  The time period between entering the recovery room amd discharge from recovery room
Incidence of postoperative residual neuromuscular blockade (rNMB) | After operation within 24 hours
  Incidence of postoperative residual neuromuscular blockade (rNMB) (defined as a train-of-four ratio, TOFR <0.9) measured 30 min after administration of the reversal agent.
The incidence of adverse effects | Within 48 hours after operation
  Unit: %; This value is a percentage. Any adverse effects in the operating room or in PACU include procedural pain, nausea, vomiting, dizziness, pruritus, reintubation, incision site complication, postprocedural nausea, vomiting, flatulence, procedural complication, insomnia, muscular weakness, headache, pharyngolaryngeal pain.
Number of patients who need rescue medication | After operation within 24 hours
  After extubation to prior to discharge from the recovery room, record the number of patients who need rescue medication because of clinical signs of residual paralysis (i.e. if a patient complain about muscle weakness, difficulty breathing, or oxygen desaturation ≤ 95%)
The incidence of mean arterial blood pressure fluctuations ≥20% | After operation within 24 hours
  The proportion of patients in this group who experience mean arterial blood pressure fluctuation ≥ 20% within 30 minutes after administration of antagonists compared with before administration of antagonists
The incidence of heart rate fluctuations ≥20% | After operation within 24 hours
  The proportion of patients in this group who experience heart rate fluctuation ≥ 20% within 30 minutes after administration of antagonists compared with before administration of antagonists
The incidence of postoperative pulmonary complications | Within the first 7 days after surgery
  Unit: %; This value is a percentage. Postoperative pulmonary complications include pneumonia; aspiration pneumonitis; atelectasis; respiratory failure; bronchospasm; pulmonary congestion; pleural effusion; pneumothorax.
Unplanned ICU hospitalization rate | 1 months after operation
  Unit: %; This value is a percentage.
Hypoxemic events | participants will be followed for the duration of the PACU stay, an expected average of 2 hours, up to 7 days
  Blood oxygenation values will be measured using pulse oximetry from the time of PACU admission until discharge from the PACU

CONTACTS AND LOCATIONS:
Overall Officials: Guyan Wang, Study Director — Beijing Tongren Hospital
Locations (2):
- China (2):
  - Beijing tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cata JP, Lasala JD, Williams W, Mena GE. Myasthenia Gravis and Thymoma Surgery: A Clinical Update for the Cardiothoracic Anesthesiologist. J Cardiothorac Vasc Anesth. 2019 Sep;33(9):2537-2545. doi: 10.1053/j.jvca.2018.07.036. Epub 2018 Jul 29. PMID 30219643
- [Background] Sheikh S, Alvi U, Soliven B, Rezania K. Drugs That Induce or Cause Deterioration of Myasthenia Gravis: An Update. J Clin Med. 2021 Apr 6;10(7):1537. doi: 10.3390/jcm10071537. PMID 33917535
- [Background] Vymazal T, Krecmerova M, Bicek V, Lischke R. Feasibility of full and rapid neuromuscular blockade recovery with sugammadex in myasthenia gravis patients undergoing surgery - a series of 117 cases. Ther Clin Risk Manag. 2015 Oct 15;11:1593-6. doi: 10.2147/TCRM.S93009. eCollection 2015. PMID 26508869
- [Background] van den Bersselaar LR, Gubbels M, Riazi S, Heytens L, Jungbluth H, Voermans NC, Snoeck MMJ. Mapping the current evidence on the anesthetic management of adult patients with neuromuscular disorders-a scoping review. Can J Anaesth. 2022 Jun;69(6):756-773. doi: 10.1007/s12630-022-02230-3. Epub 2022 Mar 23. PMID 35322378
- [Background] Fernandes HDS, Ximenes JLS, Nunes DI, Ashmawi HA, Vieira JE. Failure of reversion of neuromuscular block with sugammadex in patient with myasthenia gravis: case report and brief review of literature. BMC Anesthesiol. 2019 Aug 17;19(1):160. doi: 10.1186/s12871-019-0829-0. PMID 31421671
- [Background] No HJ, Yoo YC, Oh YJ, Lee HS, Jeon S, Kweon KH, Kim NY. Comparison between Sugammadex and Neostigmine after Video-Assisted Thoracoscopic Surgery-Thymectomy in Patients with Myasthenia Gravis: A Single-Center Retrospective Exploratory Analysis. J Pers Med. 2023 Sep 15;13(9):1380. doi: 10.3390/jpm13091380. PMID 37763148
- [Background] Schaller SJ, Lewald H. Clinical pharmacology and efficacy of sugammadex in the reversal of neuromuscular blockade. Expert Opin Drug Metab Toxicol. 2016 Sep;12(9):1097-108. doi: 10.1080/17425255.2016.1215426. Epub 2016 Aug 3. PMID 27463265
- [Background] Tsukada S, Shimizu S, Fushimi K. Rocuronium reversed with sugammadex for thymectomy in myasthenia gravis: A retrospective analysis of complications from Japan. Eur J Anaesthesiol. 2021 Aug 1;38(8):850-855. doi: 10.1097/EJA.0000000000001500. PMID 34226417
- [Background] de Boer HD, Shields MO, Booij LH. Reversal of neuromuscular blockade with sugammadex in patients with myasthenia gravis: a case series of 21 patients and review of the literature. Eur J Anaesthesiol. 2014 Dec;31(12):715-21. doi: 10.1097/EJA.0000000000000153. No abstract available. PMID 25192270
- [Background] Mouri H, Jo T, Matsui H, Fushimi K, Yasunaga H. Effect of Sugammadex on Postoperative Myasthenic Crisis in Myasthenia Gravis Patients: Propensity Score Analysis of a Japanese Nationwide Database. Anesth Analg. 2020 Feb;130(2):367-373. doi: 10.1213/ANE.0000000000004239. PMID 31124838
- [Background] Fujimoto M, Terasaki S, Nishi M, Yamamoto T. Response to rocuronium and its determinants in patients with myasthenia gravis: A case-control study. Eur J Anaesthesiol. 2015 Oct;32(10):672-80. doi: 10.1097/EJA.0000000000000257. PMID 26086278
- [Background] Lai HC, Huang TW, Tseng WC, Wu TS, Wu ZF. Sugammadex and postoperative myasthenic crisis. J Clin Anesth. 2019 Nov;57:63. doi: 10.1016/j.jclinane.2019.02.026. Epub 2019 Mar 12. No abstract available. PMID 30875518
- [Background] Keating GM. Sugammadex: A Review of Neuromuscular Blockade Reversal. Drugs. 2016 Jul;76(10):1041-52. doi: 10.1007/s40265-016-0604-1. PMID 27324403
- [Background] Petrun AM, Mekis D, Kamenik M. Successful use of rocuronium and sugammadex in a patient with myasthenia. Eur J Anaesthesiol. 2010 Oct;27(10):917-8. doi: 10.1097/EJA.0b013e3283392593. No abstract available. PMID 20375901
- [Background] Kiss G, Lacour A, d'Hollander A. Fade of train-of-four ratio despite administration of more than 12 mg kg(-1) sugammadex in a myasthenia gravis patient receiving rocuronium. Br J Anaesth. 2013 May;110(5):854-5. doi: 10.1093/bja/aet098. No abstract available. PMID 23599531
- [Background] Gurunathan U, Kunju SM, Stanton LML. Use of sugammadex in patients with neuromuscular disorders: a systematic review of case reports. BMC Anesthesiol. 2019 Nov 19;19(1):213. doi: 10.1186/s12871-019-0887-3. PMID 31744470
- [Background] Jones RK, Caldwell JE, Brull SJ, Soto RG. Reversal of profound rocuronium-induced blockade with sugammadex: a randomized comparison with neostigmine. Anesthesiology. 2008 Nov;109(5):816-24. doi: 10.1097/ALN.0b013e31818a3fee. PMID 18946293
- [Background] Blobner M, Eriksson LI, Scholz J, Motsch J, Della Rocca G, Prins ME. Reversal of rocuronium-induced neuromuscular blockade with sugammadex compared with neostigmine during sevoflurane anaesthesia: results of a randomised, controlled trial. Eur J Anaesthesiol. 2010 Oct;27(10):874-81. doi: 10.1097/EJA.0b013e32833d56b7. PMID 20683334
- [Background] Suy K, Morias K, Cammu G, Hans P, van Duijnhoven WG, Heeringa M, Demeyer I. Effective reversal of moderate rocuronium- or vecuronium-induced neuromuscular block with sugammadex, a selective relaxant binding agent. Anesthesiology. 2007 Feb;106(2):283-8. doi: 10.1097/00000542-200702000-00016. PMID 17264722
- [Background] Reid JE, Breslin DS, Mirakhur RK, Hayes AH. Neostigmine antagonism of rocuronium block during anesthesia with sevoflurane, isoflurane or propofol. Can J Anaesth. 2001 Apr;48(4):351-5. doi: 10.1007/BF03014962. PMID 11339776